CLINICAL TRIAL: NCT01364701
Title: A Prospective, Randomized, 3-arm Parallel Trial to Evaluate the Safety and Clinical Effectiveness of 2 Lower Dose Combined PDE5i's vs. Single Maximal Dose PDE5i Treatment
Brief Title: Evaluation of Safety and Effectiveness of 2 Lower Dose Combined PDE5i's Versus Single Maximal Dose PDE5i Treatment
Acronym: PDE5i
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Ilan Gruenwald MD, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0449-10-RMB
Record Dates: First submitted 2011-05-18; First posted 2011-06-02 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-04

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; combination therapy; Sildenafil; tadalafil; PDE5i; No Conditions
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Maximal dose sildenafil (Active Comparator): 4 tablets of sildenafil 100mg are given for on demand use
  Interventions: Drug: Sildenafil 100 mg
- Tadalafil 20mg maximal dose (Active Comparator): 4 tablets of tadalafil 20mg are given for on demand use
  Interventions: Drug: Tadalafil 20 mg
- Combination half dose (Active Comparator): 4 tablets of sildenafil 50mg and tadalafil 10mg are given for on demand use
  Interventions: Drug: Combination half of maximal dose for sildenafil & tadalafil

INTERVENTIONS:
Drug: Sildenafil 100 mg — 4 tablets for on demand use
  Other Names: Viagra
  Arms: Maximal dose sildenafil
Drug: Tadalafil 20 mg — 4 tablets on demand
  Other Names: Cialis
  Arms: Tadalafil 20mg maximal dose
Drug: Combination half of maximal dose for sildenafil & tadalafil — 4 tablets on demand
  Other Names: Combination
  Arms: Combination half dose

SUMMARY:
Clinical effectiveness is of the finest tools to evaluate treatment success and is combined of 3 elements: treatment effectivity, side effect profile and patient compliance. Since the 3 main PDE5i's differ in their molecular structure, therapeutic profile and pharmacokinetics, it seems logical to assume that combining 2 different PDE5i's at lower dosage each may be beneficial in comparison to a single PDE5i maximal dose therapy. The aim of this study is to compare the clinical effectiveness of combination therapy (2 lower-dose PDE5i's) versus single maximal dose PDE5i therapy.

DETAILED DESCRIPTION:
This will be a prospective, randomized, 3-arm parallel trial on 60 males with erectile dysfunction (ED) that have never been exposed to PDE5i therapy (naïve patients) will be enrolled. In each group, every patient will receive three treatment regimes (Viagra®50mg & Cialis®10mg, Viagra®100mg, Cialis®20mg), in different sequences of administration.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging between 35-75 years.
* Sexually active
* IIEF ED domain score 22 and below

Exclusion Criteria:

* Subjects with premature ejaculation as their main sexual complaint.
* Subjects with severe cardiovascular disease
* Subjects with Contraindications to PDE5i therapy. Namely patients receiving treatment with nitrate based medication or patients that for various reasons cannot take PDE5 inhibitors (i.e severe coronary disease, liver or renal failure, concomitant medications, etc.).

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function-Erectile Dysfunction (IIEF-ED) Domain Score | Every visit- altogether 3 months
  At each visit after use of different treatment each time

SECONDARY OUTCOMES:
Erection Hardness Scale | Each visit- altogether 3 months
  At each visit after use of different treatment each time

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Vardi, Prof., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel